CLINICAL TRIAL: NCT04313946
Title: The Benefits of Artificial Intelligence Algorithms (CNNs) for Discriminating Between COVID-19 and Influenza Pneumonitis in an Emergency Department Using Chest X-Ray Examinations
Brief Title: Artificial Intelligence Algorithms for Discriminating Between COVID-19 and Influenza Pneumonitis Using Chest X-Rays
Acronym: AI-COVID-Xr
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Professor Adrian Covic (Other)
Collaborators: Falcon Trading Iasi (Unknown); Romanian Academy of Medical Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Professor Adrian Covic, Clinical Professor, Grigore T. Popa University of Medicine and Pharmacy
Organization: Grigore T. Popa University of Medicine and Pharmacy (Other)
Other Study IDs: 0110
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Pneumonia, Viral; Influenza With Pneumonia; Flu Symptom; Flu Like Illness; Pneumonia, Interstitial; Pneumonia, Ventilator-Associated; Pneumonia Atypical
Keywords: Artificial Intelligence; CNNs; COVID-19; chest X-Ray; Emergency Department; Triage; Flu
MeSH Terms: conditions — COVID-19; Pneumonia, Viral; Lung Diseases, Interstitial; Pneumonia, Ventilator-Associated; Pneumonia, Mycoplasma; Emergencies; Influenza, Human

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic Patients: Our goal is to identify an artificial intelligence algorithm that can be run on lung radiographs in patients with influenza / respiratory viral symptoms who come to the emergency department / triage. This algorithm aims to identify the radiographs of patients with COVID-19 and those with influenza pneumonitis, with accuracy verified by COVID-19 tests.
  Interventions: Diagnostic Test: Scanning Chest X-rays and performing AI algorithms on images

INTERVENTIONS:
Diagnostic Test: Scanning Chest X-rays and performing AI algorithms on images — Chest X-Rays; AI CNNs; Results

SUMMARY:
This project aims to use artificial intelligence (image discrimination) algorithms, specifically convolutional neural networks (CNNs) for scanning chest radiographs in the emergency department (triage) in patients with suspected respiratory symptoms (fever, cough, myalgia) of coronavirus infection COVID 19. The objective is to create and validate a software solution that discriminates on the basis of the chest x-ray between Covid-19 pneumonitis and influenza

DETAILED DESCRIPTION:
This project aims to use artificial intelligence (image discrimination) algorithms;

* specifically convolutional neural networks (CNNs) for scanning chest radiographs in the emergency department (triage) in patients with suspected respiratory symptoms (fever, cough, myalgia) of coronavirus infection COVID 19;
* the objective is to create and validate a software solution that discriminates on the basis of the chest x-ray between Covid-19 pneumonitis and influenza;
* this software will be trained by introducing X-Rays from patients with/without COVID-19 pneumonitis and/or flu pneumonitis;
* the same AI algorithm will run on future X-Ray scans for predicting possible COVID-19 pneumonitis

ELIGIBILITY:
Inclusion Criteria:

* flu-like symptoms: myalgia, cough, fever, sputum
* Chest X-Rays
* COVID-19 biological tests

Exclusion Criteria:

* patient refusal
* uncertain radiographs
* uncertain tests results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with influenza symptoms that arrive at emergency department with cough, fever, myalgia - which are suspected of COVID-19 infection
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-08-16 (Estimated); Study Completion 2020-08-18 (Estimated)

PRIMARY OUTCOMES:
COVID-19 positive X-Rays | 6 months
  Number of participants with pneumonitis on Chest X-Ray and COVID 19 positive
COVID-19 negative X-Rays | 6 months
  Number of participants with pneumonitis on Chest X-Ray and COVID 19 negative

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Burlacu, Lecturer, Principal Investigator — University of Medicine and Pharmacy Gr T Popa - Iasi; Radu Dabija, Lecturer, Principal Investigator — University of Medicine and Pharmacy Gr T Popa - Iasi
Locations (3):
- U.O. Multidisciplinare di Patologia Mammaria e Ricerca Traslazionale; Dipartimento Universitario Clinico di Scienze Mediche, Chirurgiche e della Salute Università degli Studi di Trieste, Cremona, Italy
- University of Medicine and Pharmacy Gr T Popa, Iași, Romania
- Department of Cardiology at Chelsea and Westminster NHS hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Yes, we would be happy to share the algorithm code and the results with any scientist interested (without any financial interests)
Supporting Information: Study Protocol, ICF, Analytic Code